CLINICAL TRIAL: NCT03896828
Title: Practical Approaches for Interrupting Prolonged Sitting to Improve Postprandial Glucose and Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SSW
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Fourteen men and women will visit the lab on three separate occasions and will remain seated at a desk all-day (Visit 1) or interrupt this sitting every 30-minutes with either 2-minute walking-breaks (Visit 2) or with 15 body-weight squats (repeatedly rising from a chair and onto tip-toes, Visit 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sedentary (Experimental): Sedentary (SED): Participants will remain seated in the lab all-day (7.5 hr).
  Interventions: Dietary Supplement: Mixed-macronutrient meal
- Walking Breaks (Experimental): Walking breaks (WALK): Participants will perform 2-minute walking breaks at 3.1 mph on a treadmill every 30 minutes (7.5 hr).
  Interventions: Dietary Supplement: Mixed-macronutrient meal
- Resistance-exercise breaks (Experimental): Resistance exercise breaks (RE): Participants will perform 15 "squats" (1-minute) every 30 minutes. To reduce the risk of injury, standardize squat-depth, and recruit similar muscle groups as walking, the squats performed will be a "chair-stand with calf-raise" (7.5 hr).
  Interventions: Dietary Supplement: Mixed-macronutrient meal

INTERVENTIONS:
Dietary Supplement: Mixed-macronutrient meal — Participants will be provided a mixed-macronutrient meal (liquid drink) at hours "0" and "3", mimicking the energy and macronutrient composition of breakfast and lunch in Western society (38). 20% of daily energy intake will be provided as "breakfast" and 30% at lunch. Macronutrient composition will reflect a diet providing 55% energy needs from carbohydrate (CHO) and 1.2g/kg/d protein. The remaining energy requirements, as determined by total energy intake, will be met with dietary fat (estimated to be ~0.2 and 0.3g/kg fat for breakfast and lunch, respectively), similar to previous liquid mixed-meal approaches.

SUMMARY:
The present study will determine the impact of interrupting prolonged sitting with short, 2-minute walks or body-weight squats on: i) postprandial glycemia and insulinemia, and; ii) postprandial utilization of dietary amino acids. We hypothesize that postprandial glycemia and insulinemia will be similarly improved by interrupting prolonged sitting with short walks or body-weight squats, whereas postprandial utilization of dietary amino acids will only be improved by interrupting prolonged sitting with body-weight squats.

DETAILED DESCRIPTION:
Sedentary behavior is an independent risk factor for chronic disease and premature mortality. Despite a growing awareness of the health risks associated with prolonged sitting, Americans spend upwards of 10 hours per day in a sedentary state. Many leisure-time activities and careers of modern society involve prolonged sitting, necessitating an urgent need to identify strategies that mitigate the health consequences of these behaviors. Recent evidence suggests that interrupting prolonged periods of sitting with short breaks of walking or cycling improve postprandial glucose and lipid handling throughout the day. Thus, relatively small quantities of movement represent an efficacious strategy for improving indices of metabolic health. However, more cost-effective and practical interventions that do not require extra space (i.e. walking) or equipment (i.e. cycling or a treadmill desk) beyond one's immediate sedentary space (e.g. office, desk) would help reduce real and/or perceived barriers of adopting this efficacious disease risk-reduction behavior. A currently understudied consequence of prolonged sitting may also be a desensitization of skeletal muscle's ability to use ingested protein, which overtime can result in detriments to the quantity and quality of this important tissue. Body-weight resistance exercise (RE) can augment the body's ability to use ingested protein to support the maintenance of skeletal muscle mass, and therefore may represent a novel exercise mode to minimize consequences of prolonged sitting. The proposed research will be the first to investigate the influence of interrupting prolonged sitting with short breaks of body-weight resistance exercise (RE) on postprandial glucose and protein metabolism. Importantly, the efficacy of this approach will be directly compared to short breaks of walking, which has previously been reported to improve postprandial glycemia in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-35 yr
* Recreationally active (≤ 150 minutes of moderate-intensity physical activity per week and no more than 3 days/week of exercise)
* VO2peak considered "good" or below based on ACSM age and sex normative values
* Experiencing regular menstrual periods and not taking hormonal oral contraceptives (females only)

Exclusion Criteria:

* Inability to perform physical activity as determined by the PAR-Q
* Inability to adhere to protocol guidelines (e.g. alcohol, standardized diet)
* Physical limitations for walking or repeatedly rising from a chair
* Regular tobacco use
* Illicit drug use (e.g. growth hormone, testosterone)
* Hormonal oral contraceptive use (females only)
* Diagnosed medical condition under the care of a physician (e.g. type 2 diabetes)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Postprandial insulin area under the curve (AUC) to breakfast and lunch | 3 hours postprandial
  The plasma insulin concentration measured by enzyme-linked immunosorbent assay area under the curve will be measured using the trapezoidal rule.

SECONDARY OUTCOMES:
Postprandial glucose area under the curve (AUC) to breakfast and lunch | 3 hours postprandial
  The plasma glucose concentration measured by hexokinase method area under the curve will be measured using the trapezoidal rule.
Skeletal muscle dietary protein incorporation | 7.5 hours postprandial
  [2H5]Phe and [13C6]Phe incorporation into new myofibrillar (contractile) proteins will be determined by LC/MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, Ph.D, Principal Investigator — University of Toronto
Locations (1):
- Goldring Center for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No